CLINICAL TRIAL: NCT03414320
Title: Proof of Concept Study for the Identification of Patient-specific Parameters for Bolus Calculators in Type 1 Diabetic Patients
Brief Title: Proof of Concept - Identification of Patient-specific Parameters for Bolus Calculators for Type 1 Diabetes
Acronym: POC-IDENTITY-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, prof dr Pieter Gillard, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BolusCalc
Record Dates: First submitted 2018-01-12; First posted 2018-01-29 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Type1 Diabetes Mellitus
Keywords: type 1 diabetes; insulin pump; bolus calculator; continuous glucose monitoring; carbohydrate to insulin ratio; insulin sensitivity factor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: proof-of-concept, open label, single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): We will gather data from this group of patients.
  Interventions: Other: Gathering data

INTERVENTIONS:
Other: Gathering data — Gathering data about sleep, heart rate, carbohydrate intake, insulin pump, continuous glucose sensor, meals.

SUMMARY:
The adoption of bolus calculators has been limited by the slow speed of the current trial and error approach. The goal of this project is to automate the determination of patient specific insulin pump parameters based on current automatic electronic logbooks of glucose measurements, carbohydrate intake, and insulin usage, by means of a mathematical model. More specifically, the investigators are interested in computing the carbohydrate to insulin ratio (CIR) and insulin sensitivity factor (ISF), which are the main parameters of bolus calculators.

The present study is a proof-of-concept, open label, single arm clinical trial to validate the new method and refine both the mathematical model and the numerical techniques in well-regulated and disciplined type 1 diabetic subject.

The study is a "trial" of the selected underlying mathematical model and the associated algorithms to simulate the glucose values of a patient with uncertain meal-data.

DETAILED DESCRIPTION:
After signing informed consent and checking eligibility criteria participants will receive uniform education related to self-monitoring of blood glucose and continuous glucose monitoring (CGM) using the CGM sensor as well as on the bolus calculator (BC). The study will take three weeks (or three sensors) per patient.

Patients should live a close to normal life and should participate in their normal daily activities. During the study, patients must consequently keep using the BC of their insulin pump, record in the insulin pump when they eat extra food outside their regular meals and when they inject extra insulin without the use of their insulin pump. Faulty 'meal markers' have to be noted in a booklet and patients will also have to take pictures of their plate for each meal or record their meals in detail in a booklet. Patients should also consequently shut off insulin delivery when they disconnect their insulin pump and write it down in a booklet. The patients will be asked to wear an activity tracker (i.e. Fitbit), this data will help in the refinement of the model and will be used for research later in the same project.

During the study, patients must skip a total of three meals: breakfast, lunch and dinner (not on the same day, but within the three weeks). This gives the investigators a period of measurements in which they know that there are no significant amounts of unpredictable carbohydrates in the blood. Patients can give correction insulin or take extra fast carbohydrates to correct the glycaemia when needed and record this in the insulin pump or in a booklet. The fast rescue carbohydrates should be in the form of Dextro energy tablets (provided by the study team).

After the three weeks, patients will come back to the hospital where the study team will download data from the insulin pump, CGM sensor, and activity tracker. The booklet and photographs of the meals will be handed over to the study team. This is the end of the study for the patient. The collected patient data will further be used to assess the model fit of the chosen mathematical model as in, i.e. the investigators evaluate how well the model is able to reproduce the collected data.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patient followed at the endocrinology department of UZ Leuven
* Type 1 diabetes
* Treated with subcutaneous insulin pump (CSII) for more than 12 weeks
* Using a continuous glucose monitor (CGM) for more than 12 weeks
* No known diabetic gastroparesis
* C-peptide negative
* HbA1c between 6-10%
* Using, or willing to use, the bolus calculator

Exclusion Criteria:

* Type 2 diabetes, patients with secondary diabetes
* Patients treated with multiple daily insulin injections or begin of treatment with CSII less than 12 weeks before inclusion
* Known diabetic gastroparesis
* C-peptide positive
* HbA1c < 6% or > 10%
* Not using or not willing to use the bolus calculator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Accepting mathematical model | three weeks
  The primary outcome measure will be to accept or reject the mathematical model by calculating mean-squared error differences with the data.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided